CLINICAL TRIAL: NCT05815589
Title: Prosthetic Maintenance Assessment For Implant Fixed Complete Dentures With Implant Overdentures. A Randomized Clinical Trial
Brief Title: Maintenance Assessment For Implant Fixed Complete Dentures With Implant Overdentures. A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed awaad, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31922.
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Complications Implants
Keywords: Dental Prosthesis, Implant-Supported*, Denture, Overlay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): screw retained prosthesis group this group will received a mandibular screw retained hybrid prosthesis over four inra-foraminal implant
  Interventions: Other: screw retained prosthesis group
- active comparator (Active Comparator): this group received a mandibular telescopic attached overdenture.
  Interventions: Other: screw retained prosthesis group

INTERVENTIONS:
Other: screw retained prosthesis group — hybrid prosthesis screwed on four mandibular intra-foraminal implants
  Other Names: hybrid prosthesis

SUMMARY:
There are two types of complications in implant prosthesis: biologic and prosthetic . Biologic complications refer to disorders in implant function that disturb the supporting peri-implant tissues resulting in mucositis or periimplantitis in severe conditions, the technical complications refer to subjecting the implant, implant parts and /or the superstructures to a damage ,such as screw loosening ,attachment wear, fracture to part of the prosthesis or some of its teeth. Prosthetic complications after the insertion of the final prosthesis may or may not lead to implant loss but lead to an increase demand for repair and maintenance.

This study aimed to assess whether the telescopic overdenture as a removable prosthesis would necessitate maintaince at frequency similar to that with screw retained hybrid overdenture as a fixed prosthesis.

DETAILED DESCRIPTION:
Sample size calculation This power analysis used frequency of implant complications as the primary outcome. Based upon the results of Ragheb NA et al (2021) [15];the proportions of complications were 0.407 and 0.037 in the two groups, respectively. Using alpha (α) level of (5%) and Beta (β) level of (20%) i.e., power = 80%; the minimum estimated sample size was 19 implants per group. Sample size was increased to twenty-two implants per group to compensate for a drop-out rate of 30% after two years. Sample size calculation was performed using G*Power Version 3.1.9.2.

Patients were recruited in the study from the Outpatient Clinic of the Prosthodontics Department, Faculty of Dentistry, Cairo University. All of which were dissatisfied from their previous denture experience and seeking better retention to their mandibular denture. Patients had received verbal and written information about the study procedures and a written informed consent was signed prior to participation.

This study is a randomized clinical trial which was approved by the Ethics Committee of Scientific Research of Cairo University.

In this study , all participants had to install four interforaminal implants to receive either telescopic over-denture or screw retained denture.

Before the prosthetic phase, both groups were randomly assigned according to a computerized random allocation program where data of randomization were entered by the secretary of the department who neither participated in recruitment nor in examination procedures.

Randomization and Allocation concealment was guaranteed as the randomization table was locked with the study coordinator who wasn't involved in any clinical intervention. operator was informed about the treatment modality in a sealed enveloped delivered by the secretary of the department before impression procedures.

Data collection was done by the study coordinator , Blinding of the operator or data collector was not applicable due to the clear difference between the two prostheses but collected data was coded prior to sending to the statistician (blinded statistician).

A preoperative CBCT scan was taken for the participant 's mandibular arch with a scan appliance .The surgical steps were explained for all the participants and an informed consent was signed before surgery.

Intra-foraminal root form tapered threaded dental implants (Neo Biotech Co. Ltd, Seoul, Korea) were installed with 3.5/ 11.5 mm for the anterior and 3.5/10 mm for posterior sites .

Three months later, the surgical stent was used to relocate the implants position for uncovering and the healing abutment was screwed with collar height 5mm to allow for proper gingival healing around the implants prior making the impression.

The impression was made with an open tray splinted implant level impression technique According to randomization, either a telescopic implant supported overdenture or a screw retained denture was fabricated for each case.

During the follow -up period, prosthetic complications were grouped and their frequency was documented according to the type of prosthesis . Both prosthetic and biological aspects were included.

Each complication was documented with stating the frequency of its occurrence, any complication was managed and repaired.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous male patients between the age of 50-70 years. patients with HB=bA1C up to 8 with normal blood sugar (79-110) Sufficient bone width (≥ 6 mm) It could be either normally present or achieved by bone plateauing. This will be confirmed by cone beam computed tomographic (CBCT) scans.

Residual bone height ranging from 11-15 mm Patients seeking to install implant and for whom new dentures will be constructed.

Patients, who are dissatisfied with the retention and stability of their technically satisfactory dentures.

Patients providing written informed consents to participate in the trial and this will be done before the scheduled date for implant installation.

Exclusion Criteria:

Any systemic disease that may interfere with dental implants placement and/or Osseointegration as; uncontrolled diabetes, hypertension, osteoporosis and irradiation. Heavy smoker (more than 20 cigarette / day) Patients with parafuctional habits as bruxism and clenching

-

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients were selected to avoid female hormonal changes, calcium insufficiency and osteoporosis which have a high prevalence among females which may affect the Osseointegration of placed implants.
Enrollment: 44 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Maintenance | one year
  maintenance for complication assed through counting frequency of incidence

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Elkady phd, Study Director — lecturer
Locations (3):
- Egypt (3):
  - Cairo university, Cairo
  - Doaa Mahmoud Elkady, Cairo
  - Nesma Mohamed Awaad, Cairo

IPD SHARING:
Plan to Share IPD: No